CLINICAL TRIAL: NCT02682472
Title: SettleIN - An Adjustment to Care Intervention for People With Dementia: A Feasibility Pilot Study in Care Homes
Brief Title: SettleIN - Adjustment to Care in Dementia: An Intervention Feasibility Study v0.1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15/0201; 15/LO/0611 (Other: NRES Committee London - Camden & Kings Cross)
Record Dates: First submitted 2016-01-22; First posted 2016-02-15 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SettleIN (Experimental): SettleIN - Adjustment to care programme intervention
  Interventions: Other: SettleIN - Adjustment to care programme

INTERVENTIONS:
Other: SettleIN - Adjustment to care programme — A programme for care home staff to support new residents with dementia quickly and successfully adjust to life in a care home

SUMMARY:
Admission into a care home for people with dementia has been linked with both positive and negative psychological outcomes for both the resident and their carers. Whilst some people with dementia adjust quickly, many never adjust at all or adjustment is complex and linked to cognitive and behavioural decline (Wilson et al, 2007). Therefore, support for healthy adjustment is needed.

Recent research (Aminzadeh et al., 2013; Sury, Burns and Brodaty, 2013, Sussman and Dupuis, 2013) has identified factors that influence different relocation outcomes and prevent adverse reactions. There are currently no interventions that support successful adjustment by emphasising the positive factors found to influence relocation outcomes while mitigating the effects of negative influences and addressing any missed pre-admission procedures, reported in the literature.

The current project seeks to design an intervention that predominantly builds on the work of Sury et al (2013) and focuses on promoting healthy adjustment through an enhanced best practice based admission process.

The intervention will be developed through systematic review of the literature and consultation with professional experts, service users, care home staff and carers. The current study will serve as a feasibility (pilot) study and test the acceptability of the intervention design, examine recruitment and dropout and establish sample size for future, larger studies. It also aims to examine whether the intervention indicates an improvement in residents' quality of life, mood, overall adjustment and carer satisfaction with care.

All participants will receive a subset of the same intervention, specifically tailored to their needs and with elements delivered by staff, carer or psychologist. Staff and researchers will assess the improvement indicators mentioned above using relevant psychometric measures at baseline, post intervention completion and at one-month follow up. Indirect measures (interviews and staff field notes) will also be used to indicate intervention fidelity and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Site:

  * Within Greater London
  * At least one resident who has been recently admitted to care (ideally within the previous fortnight and no more than one month after admission).
  * Sufficient cover to allow at least 1 staff lead to attend a half-day training
  * Managerial assurance of adequate resources allowing staff participation

Resident sample:

* Meet diagnostic criteria for dementia according to the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V, APA, 2013)
* Score between FAST stage 2 and 6 representing a range of mild to moderately severe dementia on The Functional Assessment Staging Test (FAST, Reisberg, 1987)
* Be able to communicate in English

Staff sample:

• Working as a Nurse (registered nurses of any grade, student nurses) or Care Assistant (Health Care Assistants and nursing assistants).

DSM Criteria will be confirmed by formal diagnosis or use of the FAST as a screen.

Exclusion Criteria:

Site:

• Participation in any other research study

Resident sample:

• Score FAST stage 7 equating to severe dementia on The Functional Assessment Staging Test (FAST, Reisberg, 1987)

Staff sample:

• Lack of availability on training, intervention delivery and assessment dates

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-07-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is change in residents' quality of life and measured by the Quality of Life in Alzheimer's Disease (QOL-AD, Lodgson et al, 1996) which will be administered by researchers. | Baseline, post intervention (4-6 weeks after intervention start) and at one month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Spector, Principal Investigator — UCL London
Locations (1):
- Multiple UK Care Home locations, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised and summarised data is planned for inclusion in an empirical paper to be submitted for publication. The summarised results will be fed back to participating care home managers and staff if desired.